CLINICAL TRIAL: NCT01608256
Title: Assessing the Effect of MCI on Driving Ability by Using on Road Driving Test. The Relationship Between Their Driving Outcome and Their Cognitive Decline Will be Examined
Brief Title: Driving Ability Among People With Mild Cognitive Impairment
Acronym: MCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Areej Wishahi, Student for the MA degree, Tel Aviv University
Other Study IDs: ק0012012
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; Automobile Driving; cognitive aspects
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mild cognitive impairment: men and women, aged 50 to 70. The inclusion criteria are:diagnosis of MCI (given by a neurologist), valid driver's license and driving experience of at least a year. the exclusion criteria are: people diagnosed with other neurological damage such as: dementia, CVA and head injury, people with sensory or motor impairment.
- Healthy people: Men and women, ages 50-70. the inclusion criteria are: healthy people with out neurological disease or psychiatric illness, have valid driver's license and driving experience of at least a year.

SUMMARY:
The Purpose of this study is to assess the effect of MCI on driving ability by using on road driving test. The relationship between their driving outcome and their cognitive decline will be examined.

DETAILED DESCRIPTION:
Each subject will be evaluated by test battery which is accepted to driving assessment and include: The Montreal Cognitive Assessment, Clock Drawing Task, Color Trail Test, Motor Free Visual Perception, Visual Spatial Search Task , Awareness Questionnaire and on road driving test.

The difference between outcome measures of the on road test between the patient group and the control group will be tested. The correlation between outcome measures of the on road test and the cognitive tests will be examined.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment(given by a neurologist), valid driver's license and driving experience of at least a year.

Exclusion Criteria:

* people diagnosed with other neurological damage such as: dementia, CVA and head injury, people with sensory or motor impairment

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-07 (Estimated); Study Completion 2014-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sherotw breot Clalit, Hedera, Israel